CLINICAL TRIAL: NCT02661230
Title: Design of a Cognitive Motor Intervention Using a Video Game to Enhance Brain Activity: A Feasibility Study Including Healthy Participants and Heart Patients on the Intensive Care Unit
Brief Title: Virtual Reality Exercise on the Intensive Care Unit in Heart Patients
Acronym: VRICUGAMING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VRICU-Study
Record Dates: First submitted 2016-01-11; First posted 2016-01-22 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Motor Activity
Keywords: exergaming; intensive care unit; feasibility acceptability; heart; brain function
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- COGNIPLUS (Experimental): Exercise-Gaming
  Interventions: Device: COGNIPLUS

INTERVENTIONS:
Device: COGNIPLUS — Run 1 Video game: Phasic Alertness (Alert S1) Instruction phase 2 minutes, 2 x 3 minutes of rest, followed by 5 x 60 sec of video game activity, alternating with 60 sec of rest.
  Run 2 Video game: Intrinsic Alertness (Alert S2) Instruction phase 2 minutes, 2 x 3 minutes of rest, followed by 5 x 60 sec of video game activity, alternating with 60 sec of rest.
  Run 3 Video game: Visual modality (Select S1) Instruction phase 2 minutes, 2 x 3 minutes of rest, followed by 5 x 60 sec of video game activity, alternating with 60 sec of rest.
  Run 4 Video game: Acoustic / Stimulus Combinations (Select S2) Instruction phase 2 minutes, 2 x 3 minutes of rest, followed by 5 x 60 sec of video game activity, alternating with 60 sec of rest.

SUMMARY:
This project proposes the development and design of a motor intervention using a cognitive video game and describes the feasibility, safety and acceptability of virtual augmented video gaming device named Virtual Reality on the Intensive Care Unit (VRICU). The project in two phases is performed in healthy participants (Phase 1) and heart patients after elective heart surgery on the Intensive Care Unit (Phase 2).

Furthermore, brain function will be measured during exer-gaming with the VRICU device with non-invasive instruments (fNIRS/EEG) in both the healthy participants and the heart patients.

The VRICU device is a patient friendly construction to allow a patient exergaming in bed. The project is a cooperation between scientist at the USZ (physiotherapist / anaesthsiologists / engineers), human movement scientist at the ETHZ and (poly- / electro-) mechanics at the Paul Scherrer Institut.

DETAILED DESCRIPTION:
There is converging evidence at systems levels that physical exercise participation is beneficial to cognition, especially to the different subtypes of attention. Such evidence highlights the importance of promoting physical exercise to prevent or reverse cognitive and neural decline. Accordingly, physical exercise can serve to promote function in patients. Physical exercise games may be engaged to gauge performance increases in motor learning and early rehabilitation programs as performed on an intensive care unit.

This project proposes the development and design of a cognitive motor intervention using a custom video game (which will be performed in supine position in bed) to enhance brain activity and describes the feasibility, safety and acceptability of virtual augmented video dance gaming.

This project is divided in two (2) phases:

Phase1 The patients are not expected to exercise the video game in the usual standing position due to their condition. Thus, we designed a patient friendly construction with colleagues of the construction department of the Paul Scherrer Institute (Villigen, Switzerland), which enables video game exercising in supine position. This construction and custom video game will be tested first in healthy participants for feasibility, acceptability and safety. Furthermore, brain activity of the participants will be measured and evaluated, before during and shortly after playing the video game in 15 healthy participants.

Phase 2 After the device and procedures tested in phase 1 is feasible, acceptable and safe, maximal 10 patients on the ICU ward (receiving elective heart surgery, will be recruited to evaluate the feasibility, safety, acceptability and effect on brain function of a custom video exercise game.

The aims of this study are:

Phase 1 Objective To determine the feasibility, safety acceptability and effect of brain function of a cognitive motor intervention using a custom video game in healthy participants.

Phase 2 Objectives To determine the feasibility, safety and acceptability (if possible) of a cognitive motor intervention using a custom video game at the Intensive Care Unit.

Evaluation of brain functions before, during and after exercising using a video game.

ELIGIBILITY:
Inclusion Criteria:

Phase 1

Healthy participants

* 18 years or older of age.
* In good health and not under treatment of a physician

Phase 2

Patient on the intensive care unit. Inclusion criteria

* Adult patients (>18 years).
* Signed informed consent by patient.
* Patient awake and close to full cooperation needed to Participate actively in the experimental intervention.

Exclusion Criteria:

Phase 1

• No exclusion criteria

Phase 2

Exclusion criteria for the patients are:

* Known epilepsy
* Inability to obtain consent
* known or suspected non-compliance
* raised intracranial pressure
* participation in conflicting study
* known dementia
* absence of a limb
* Sepsis
* Incapable of discernment -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Feasibility & usibility 1 | Healthy participants 120 minutes, patients: dependent on physical ability
  Intensity: Level of gameplay
Feasibility & usibility 2 Feasibility & Usibility 2 | Healthy participants 120 minutes, patients: dependent on physical ability
  Accuracy: Percentage
Feasibility & usibility 3 | Healthy participants 120 minutes, patients: dependent on physical ability
  Time: Minutes

SECONDARY OUTCOMES:
Safety parameters & adverse effects of the VRICU device | Minimal 1 up to 30 Minutes (if applicable)
  Assessment of (Serious) Adverse Events and Other Safety Related Events An unexpected SAE refers to any AE, the nature or severity of which is not consistent with the applicable product information, namely please specify for unapproved investigational medicinal products the current Investigator's Brochure and the approved instructions for devices with CE-marking.
  The investigator will promptly review documented AEs and abnormal test findings to determine
  * if the abnormal test finding should be classified as an AE,
  * if there is a reasonable possibility that the AE was caused by the investigational device or study treatment(s), and
  * if the AE meets the criteria for an SAE.
MOSRAM Questionnaire | 10 minutes
  Participant & Patient satisfactory questionnaire concerning use off technical devices and software.
functional Near Infrared Spectroscopy (fNIRS) | healthy participants 90 minutes, patients: dependent on physical ability
  fNirs outcome of frontal lobe measured in SP02%; Baseline during gameplay and during recuperation of exercise gameplay
EEG | healthy participants 90 minutes, patients: dependent on physical ability
  EEG outcome of frontal lobe during exerciseplay and recupperation measured in milliseconds

CONTACTS AND LOCATIONS:
Overall Officials: Ruud Knols, Dr., Principal Investigator — University of Zurich
Locations (1):
- Dr. Jaap Swanenburg, Zurich, Switzerland